CLINICAL TRIAL: NCT05261152
Title: Saccharomyces Boulardii in the Prevention of Antibiotic-associated Diarrhea in Hospitalized Adult Patients With Lower Respiratory Tract Infections
Brief Title: S. Boulardii in Prevention of Antibiotic-associated Diarrhea in Hospitalized Adults With Respiratory Tract Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Centre of Serbia (Other)
Collaborators: Institute for Pulmonary Diseases of Vojvodina (Unknown)
Responsible Party: Principal Investigator, Branislava Milenkovic, Prof. MD, PhD, Clinical Centre of Serbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 264/21
Record Dates: First submitted 2022-02-19; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Prevention & Control; Diarrhea Caused by Drug; Respiratory Infection Bacterial; Anti-Bacterial Agents
Keywords: Saccharomyces boulardii, antibiotic-associated diarrhea
MeSH Terms: interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Capsules are containing S. boulardii and were administered twice daily (250 mg). The administration of investigated product started within 30 min before the first dose of the antibiotic and continued for 21 days.
  Interventions: Drug: drug product: capsules are containing S. boulardii, administered twice daily (250 mg)
- Placebo group (Placebo Comparator): Capsules are containing placebo and were administered twice daily. The administration of investigated product started within 30 min before the first dose of the antibiotic and continued for 21 days.
  Interventions: Drug: drug product: capsules are containing S. boulardii, administered twice daily (250 mg)

INTERVENTIONS:
Drug: drug product: capsules are containing S. boulardii, administered twice daily (250 mg) — Randomisation: 1:1 Capsules containing S. boulardii twice daily (250 mg) or indistinguishable capsules containing placebo twice daily.
  Other Names: Sacharomyces boulardi,

SUMMARY:
Antibiotic-associated diarrhea (AAD) is the most common gastrointestinal complication of antibiotic use, with potentially serious clinical impact. The aim of this study is to assess the efficacy and safety of Saccharomyces boulardii in the prevention of AAD in adult patients with lower respiratory tract infection (LRTI) treated in a hospital.

A multicenter, randomized, parallel-group, double-blind, placebo-controlled study is conducted whereby adults who are hospitalized due to LRTI and treated with intravenous antibiotics and randomized to capsules containing S. boulardii or indistinguishable placebo. The outcome measures were: relevant clinical features, gastrointestinal symptoms, and adverse events.

DETAILED DESCRIPTION:
The participants are adult patients hospitalized due to lower respiratory tract infection (LRTI) and treated with intravenous antibiotics. They are randomized (1:1) to capsules containing S. boulardii twice daily (250 mg) or indistinguishable placebo twice daily. The administration of investigated product started within 30 min before the first dose of the antibiotic and continued for 21 days. The outcome measures (relevant clinical features, gastrointestinal symptoms, and adverse events) were assessed in 3-time points: T1 - screening, T2 - randomization, and T3 - hospital discharge.

The relevant gastrointestinal symptoms are: frequency and severity of nausea, bloating, gas production, abdominal pain, fever, stool frequency between investigated groups. The median value of stool consistency is assessed by the Bristol Stool Scale.

Visits are scheduled for V0 (screening), V1 (randomization and first use of study drug), V3 (on discharge from hospital), end of treatment (EOT) (telephone call on the 21st day after the first dose).

Inclusion criteria are: age ≥18 years, informed consent signed before joining the survey, diagnosis of LRTI, expected period of hospitalization: at least 5 days, necessity of administration of ≥5 days of intravenous antibiotics, women who have not been surgically sterilized or postmenopausal for more than a year must agree to an effective method of contraception in order to prevent conception during the research (effective methods include intrauterine devices, hormonal contraception and double protection).

Exclusion criteria are: active diarrhea, diarrhea in the previous two weeks, current therapy for C. difficile-associated diarrhea (CDAD) or active C. difficile infection and CDAD, based on the clinical picture of diarrhea with the presence of toxins A and / or B (or their genes) C. difficile in stool, number of previous CDAD episodes> 1, previously documented infection with C. difficile 8 weeks before randomization, use of broad-spectrum antibiotics for two months before the start of the study drug, antibiotics, including those not defined by the protocol for the treatment of current lower respiratory tract infection, are allowed within the first 24 hours of starting the study drug, topical treatment with a non-beta-lactam antibiotic other than a macrolide, risk of death within 90 days from the start of the study according to the investigator's clinical assessment, known hypersensitivity to the study drug or its ingredients, history of active, uncontrolled inflammatory bowel disease (Crohn's disease, ulcerative colitis, digestive tract infections (parasitic infection, Salmonella, Shigella, history of colorectal cancer, irritable bowel syndrome), aspiration pneumonia, chronic alcoholism, subjects with confirmed influenza, neutrophil count <500 cells / mm3, patients with a central vein catheter.

Aspartate Aminotransferase > 3x, Alanine Aminotransferase > 3x above the upper limit of the reference, current chemotherapy, previous organ transplantation, participation in another clinical study during the previous 30 days, inability or unwillingness to cooperate. Accordingly, the researcher should evaluate any factor (eg. other regular therapy) that may affect the validity of the treatment results.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age ≥65 years.
* Informed consent (IC) obtained and signed prior to study participation
* For female subjects: proof of being at least 1 year post-menopausal
* Expected minimum hospital stay of 5 days
* Requiring ≥5 day course of intravenous (IV) antibiotic
* Diagnosis of lower respiratory tract infection (LRTI)
* The subject is willing and able to comply with all testing and study requirements as defined in the protocol.

Exclusion Criteria:

* Active diarrhea (where diarrhea is defined as 3 or more unformed/liquid stools on day prior to randomization)
* Subjects with diarrhea in past 2 weeks
* Current treatment for CDAD or ongoing active CDAD infection, as evidenced by clinical signs of diarrhea along with the presence of toxin A and/or B (or their respective genes) of C. difficile in the stool
* Number of previous CDAD episodes >1
* Any previously documented CDI within 8 weeks prior to randomization
* Use of broad spectrum antibiotics within 2 months of start of study drug. Antibiotics including those not specified in this protocol for the treatment of the current CAP episode are allowed within 24 h of start of study drug and the protocol-defined treatment for CAP.
* Current treatment with non-beta lactam antibiotics other than macrolides
* Risk of death within 90 days of study entry according to the clinical judgment of the investigator
* Known intolerance of study drug/ingredients
* History of or active, non-controlled inflammatory bowel disease such as Crohn's Disease or ulcerative colitis; evidence of other GI infections ie parasitic infection, Salmonella, Shigella, history of colon carcinoma, irritable bowel syndrome (IBS)
* Subjects with aspiration pneumonia
* Subjects with chronic alcoholism
* Subjects with confirmed influenza
* Neutrophil count <500 cells/mm3
* Patients with subclavian central line
* AST, ALT > 3x upper limit normal (ULN)
* Active chemotherapy, receipt of organ transplant
* Participation on another clinical study within the last 30 days
* Insufficient ability or willingness to co-operate
* In the judgment of the investigator any factors (e.g. other treatment) that could invalidate the treatment result

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
gastrointestinal symptoms and signs | 21 days
  stool frequency and consistency, nausea, gas production (meteorism), bloating, abdominal pain
fever | 21 days
  symptom / measured body temperature

CONTACTS AND LOCATIONS:
Overall Officials: Branislava Milenkovic, Prof, MD, Principal Investigator — Clinic for Pulmonary Diseases, Clinical Center of Serbia
Locations (2):
- Serbia (2):
  - Clinical Center of Serbia, Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Novi Sad

IPD SHARING:
Plan to Share IPD: No